CLINICAL TRIAL: NCT07097012
Title: Concurrent Versus Sequential Administration of Tdap and RSV Vaccines in Pregnancy - A Pilot Feasibility Trial
Brief Title: Concurrent Versus Sequential Administration of Tdap and RSV Vaccines in Pregnancy
Acronym: CosTaR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Canadian Immunization Research Network (Network)
Collaborators: Ottawa Hospital Research Institute (Other); Vaccine Evaluation Center, Canada (Other); University of British Columbia (Other); Canadian Center for Vaccinology (Other); Dalhousie University (Other); IWK Health Centre (Other); Public Health Agency of Canada (PHAC) (Other Government); Centre Hospitalier Univeritaire Sainte Justine (Unknown)
Responsible Party: Principal Investigator, Bahaa Abu Raya, Principal Investigator, Canadian Immunization Research Network
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT25
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: RSV; Tdap - Tetanus, Diphtheria and Acellular Pertussis Vaccination; Pregnancy; Healthy
Keywords: RSV; Tdap; Pregnancy; Clinical trial; Vaccine
MeSH Terms: conditions — Diphtheria | interventions — Boostrix; Respiratory Syncytial Virus Vaccines; abrysvo; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data Safety Monitoring Board members, unless unblinding is required to provide a comprehensive safety assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Concurrent Assignment (Active Comparator)
  Interventions: Biological: Tdap Vaccine Administration; Biological: RSV Vaccine; Other: Saline (as a placebo)
- Group 2: Sequential Assignment (Active Comparator)
  Interventions: Biological: Tdap Vaccine Administration; Biological: RSV Vaccine; Other: Saline (as a placebo)

INTERVENTIONS:
Biological: Tdap Vaccine Administration — The Tdap vaccine will be administered according to the Product Monograph. Participants will be asked to look away during vaccine administration to maintain blinding.
  Other Names: BOOSTRIX; Tetanus-diphtheria-acellular pertussis
Biological: RSV Vaccine — The RSVpreF vaccine will be administered according to the Product Monograph. Participants will be asked to look away during vaccine administration to maintain blinding.
  Other Names: Respiratory syncytial virus; ABRYSVO; RSVpreF
Other: Saline (as a placebo) — Normal saline (0.5mL) will be administered as a placebo according to the Product Monograph. Participants will be asked to look away during vaccine administration to maintain blinding.
  Other Names: Normal saline

SUMMARY:
The goal of this clinical trial is to learn if the RSV vaccine (protects against respiratory syncytial virus) and Tdap vaccine (protects against pertussis) are most effective in pregnant individuals when taken together at the same visit, or separately at different visits. This clinical trial will also learn about the safety and immune responses of these vaccines in pregnancy.

The Main question:

-Is it possible to run a successful trial that tests how safe and effective it is to give Tdap and RSV vaccines in pregnancy either at the same time or one after the other, at different visits?

The Secondary question:

-To determine how safe and how well the Tdap and RSV vaccines work when given in pregnancy either at the same time or one after the other, at different visits.

The Exploratory (optional participation) questions:

* To measure the levels of antibodies against whooping cough (pertussis) and RSV in mothers at 7 and 19 months after giving birth, depending on whether they got the vaccines at the same time or one after the other during pregnancy.
* To measure whooping cough antibody levels in the babies at 2, 7, and 19 months of age, whose mothers who received the vaccines in pregnancy.
* To measure the levels of RSV antibodies in the mothers' breast milk at 1 week, 2 weeks, 4 weeks, and 2 months after giving birth.

Participants will be randomly assigned to Group 1 (vaccines given at the same time, same visit) or Group 2 (vaccines given one after the other, at different visits).

There are 4 visits as part of the main study, and 6 additional visits as part of the optional study (exploratory questions).

Visit 1-2: Blood collection and vaccines administered Visit 3-4: Blood work (cord blood sample collection from infant, after delivery, if possible) Visit 5-8: Breast milk collection Visit 8-10: Blood collection (infant blood collection only at Visit 8).

Participants will be asked to keep a diary of symptoms throughout the study.

ELIGIBILITY:
Inclusion Criteria

1. Healthy pregnant individuals with a singleton pregnancy aged 18-49 years.
2. Gestational age 28-29+6 WG at time of study screening, enrolment and randomization as per documented first trimester (less than or equal to13+6 WG) ultrasound, or the first date of last menstrual period if ultrasound not obtained in the first trimester, or the age of the embryo and the date of transfer if pregnancy resulted from assisted reproductive technology.
3. Able to comply with the study procedures required to achieve primary objective of this pilot trial (not being able to comply with procedures required to achieve exploratory objectives is not an exclusion criteria).
4. Informed consent read, understood and signed prior to study-specific procedures.

Exclusion Criteria

Any of the following:

1. Receipt of RSV vaccine anytime.
2. Receipt of immunoglobulins (except Rho D) within 1 year prior to vaccination.
3. Documented receipt of pertussis vaccine within 2 years prior to vaccination.
4. Documented pertussis infection (by culture or polymerase chain reaction) within 2 years prior to vaccination.
5. Receipt of blood transfusion products within 6 months prior to vaccination.
6. Primary or secondary immunologic disorder or immunosuppression.
7. Any conditions that, in the investigator's judgement, may interfere with subject's ability to comply with study procedures or receipt of prenatal care, such as behavioural or cognitive impairment or neuropsychiatric illness.
8. Preconception diabetes mellitus (defined as: previous diagnosis of diabetes while not pregnant OR First trimester hemoglobin A1c level of 6.5% [47.5 mmol/mol] OR First trimester fasting blood glucose 126 mg/dL [7 mmol/L]).
9. Preconception chronic hypertension (defined as: sustained elevation in the systolic blood pressure to ≥140 mmHg or the diastolic blood pressure to ≥90 mmHg, that is diagnosed either prior to pregnancy or prior to 20 WG).
10. Congenital anomalies per ultrasound.
11. Hepatitis B infection; Hepatitis C infection; Untreated syphilis.
12. Contraindication to receipt of Tdap (BOOSTRIX, GSK): a) Hypersensitivity to any component of the Tdap (BOOSTRIX, GSK) vaccine or individuals having shown signs of hypersensitivity after previous administration of diphtheria, tetanus, or pertussis vaccines; b) Encephalopathy of unknown etiology, occurring within 7 days following previous vaccination with pertussis containing vaccine; c) Transient thrombocytopenia or neurological complications following an earlier immunization against diphtheria and/or tetanus.
13. Contraindication to receipt of RSVpreF (ABRYSVOTM, Pfizer): Hypersensitivity to the active substance or to any component of the vaccine.
14. Pregnancy complications at the time of recruitment that are risk factors for preterm delivery:

    1. Gestational hypertension (defined as new onset hypertension after 20 WG of systolic blood pressure is ≥140 mmHg or the diastolic blood pressure is ≥90 mmHg on two measurements at a minimum of one hour apart);
    2. Pre-eclampsia (defined as development of gestational hypertension [as defined in #a above] and proteinuria after 20 WG (Proteinuria defined as ≥300 mg in a 24 h urine specimen, or ≥0.30 on a spot protein: creatinine ratio, or ≥1+ on a dipstick;
    3. Gestational diabetes mellitus uncontrolled at time of consent (gestational diabetes is defined as a clinical syndrome characterized by the absence of preconception diabetes mellitus [as defined in #8 above] AND identification of sustained hyperglycemia during pregnancy not due to other known causes (i.e. corticosteroids, beta-mimetics, etc.) based on positive internationally recognized oral glucose tolerance test OR fasting plasma glucose of 92-125 mg/dL [5.1-6.9 mmol/l] using venous or capillary blood samples;
    4. Fetal growth restriction (defined as estimated fetal weight below 10% using locally-accepted growth curve AND Absent or reversed end-diastolic flow of the umbilical artery Doppler OR Oligohydramnios [defined as a decreased amniotic fluid volume as defined by amniotic fluid index less than 8 cm or deepest vertical pocket less than 2 cm in the presence of intact membranes without concern for fetal anomalies contributing to its etiology]);
    5. Placenta anomalies (placenta previa and abruptio, vasa previa);
    6. Polyhydramnios (defined as abnormal increase in the volume of amniotic fluid as either a deepest vertical pocket of ≥8 cm or an amniotic fluid index of ≥24 cm);
    7. Oligohydramnios (decreased amniotic fluid volume as defined in d above);
    8. Short uterine cervix (<25 mm in the second trimester of pregnancy);
    9. A significant acute disease or oral temperature ≥38 Co within 24 hours prior to vaccination. Participants can return for evaluation to be randomized/vaccinated 72 hours after symptoms resolve, if they are still within 28-29+6 WG.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of conducting a randomized controlled trial - Screening Rate | From enrollment to the end of visit 4 (end of main study) at around 12 weeks
  To evaluate the feasibility of conducting a randomized controlled trial (RCT) that would test the safety and immunogenicity of Tdap and RSV concurrent and sequential administration in pregnancy.
  Number of participants screened monthly in each site and overall.
Feasibility of conducting a randomized controlled trial - Consent & Randomization Rate | From enrollment to the end of visit 4 (end of main study) at around 12 weeks
  To evaluate the feasibility of conducting a randomized controlled trial (RCT) that would test the safety and immunogenicity of Tdap and RSV concurrent and sequential administration in pregnancy.
  Proportion/number of participants who consent and successfully randomized out of screened individuals in each site and overall.
Feasibility of conducting a randomized controlled trial - Retention Rate | From enrollment to the end of visit 4 (end of main study) at around 12 weeks
  To evaluate the feasibility of conducting a randomized controlled trial (RCT) that would test the safety and immunogenicity of Tdap and RSV concurrent and sequential administration in pregnancy.
  Proportion of randomized participants who complete the first four study visits in each site and overall.
Feasibility of conducting a randomized controlled trial - Trial Protocol Compliance Rate | From enrollment to the end of visit 4 (end of main study) at around 12 weeks
  To evaluate the feasibility of conducting a randomized controlled trial (RCT) that would test the safety and immunogenicity of Tdap and RSV concurrent and sequential administration in pregnancy.
  Percentage of participants who do not deviate from the protocol and complete vaccination and the first four visits in each site and overall.

SECONDARY OUTCOMES:
Safety Outcomes - Rates of Adverse Events Following Immunization in Participants | Up to 14 weeks after first vaccination
  In this study, an adverse event will be categorized as an AEFI if it meets the relevant provincial reporting criteria and occurs after vaccination and up until delivery.
  Rates of Adverse Events Following Immunization in Participants.
Safety Outcomes - Rates of Adverse Events of Special Interest in Participants during Pregnancy and Delivery | Up to 14 weeks after first vaccination
  Rates of Adverse Events of Special Interest in Participants during pregnancy and delivery.
Safety Outcomes - Rates of Serious Adverse Events in Participants during Pregnancy and Delivery | Up to 14 weeks after first vaccination
  Rates of Serious Adverse Events in Participants during pregnancy and delivery.
Immunogenicity - Seroconversion rate of anti-pertussis toxin IgG | 4 weeks after vaccination with Tdap
  Seroconversion rate of anti-pertussis toxin IgG 4 weeks after vaccination with Tdap vaccine in the concurrent versus sequential groups.
  For the secondary immunogenicity outcome, fold change in antibody levels between pre-vaccination and 4-weeks after vaccination will be calculated. Seroconversion rates and their 95% CI will be calculated and described. Geometric mean concentrations of antibody levels and 95% CI will be calculated.
Immunogenicity - Seroconversion rate of anti-Filamentous hemagglutinin IgG | 4 weeks after vaccination with Tdap
  Seroconversion rate of anti-Filamentous hemagglutinin IgG 4 weeks after vaccination with Tdap vaccine in the concurrent versus sequential groups.
  For the secondary immunogenicity outcome, fold change in antibody levels between pre-vaccination and 4-weeks after vaccination will be calculated. Seroconversion rates and their 95% CI will be calculated and described. Geometric mean concentrations of antibody levels and 95% CI will be calculated.
Immunogenicity - Seroconversion rate of anti-Pertactin IgG | 4 weeks after vaccination with Tdap
  Seroconversion rate of anti-Pertactin IgG 4 weeks after vaccination with Tdap vaccine in the concurrent versus sequential groups.
  For the secondary immunogenicity outcome, fold change in antibody levels between pre-vaccination and 4-weeks after vaccination will be calculated. Seroconversion rates and their 95% CI will be calculated and described. Geometric mean concentrations of antibody levels and 95% CI will be calculated.
Immunogenicity - Seroconversion rate of Prefusion RSV F protein IgG | 4 weeks after vaccination with RSV vaccine
  Seroconversion rate of Prefusion RSV F protein IgG 4 weeks after vaccination with RSV vaccine in the concurrent versus sequential groups.
  For the secondary immunogenicity outcome, fold change in antibody levels between pre-vaccination and 4-weeks after vaccination will be calculated. Seroconversion rates and their 95% CI will be calculated and described. Geometric mean concentrations of antibody levels and 95% CI will be calculated.
Immunogenicity - Anti-Pertussis toxin IgG levels at term birth (maternal and cord sera) | Up to 14 weeks after vaccination with Tdap
  Geometric mean concentrations of antibody levels and 95% CI will be calculated.
Immunogenicity - Anti-Filamentous hemagglutinin IgG levels at term birth (maternal and cord sera) | Up to 14 weeks after vaccination with Tdap
  Geometric mean concentrations of antibody levels and 95% CI will be calculated.
Immunogenicity - Anti-Pertactin IgG levels at term birth (maternal and cord sera) | Up to 14 weeks after vaccination with Tdap
  Geometric mean concentrations of antibody levels and 95% CI will be calculated.
Immunogenicity - Prefusion RSV F protein IgG levels at term birth (maternal and cord sera) | Up to 14 weeks after vaccination with RSV vaccine
  Geometric mean concentrations of antibody levels and 95% CI will be calculated.

OTHER OUTCOMES:
(1) Exploratory: Measurement of anti-B. pertussis responses in mothers 7 and 19 months after delivery | Months 7 and 19 after delivery
  Anti-B. pertussis IgG in mothers 7 and 19 months after delivery
(1) Exploratory: Measurement of RSV antibody responses in mothers 7 and 19 months after delivery | Months 7 and 19 after delivery
  Prefusion RSV F protein IgG in mothers 7 and 19 months after delivery
(2) Exploratory: Measurement of anti-B. pertussis antibody levels in infants at 2, 7 and 19 months of age born to mothers who received concurrent and sequential administration of vaccines against pertussis and RSV in pregnancy | Infants at 2, 7 and 19 months of age
  Anti-B. pertussis IgG in infants at 2, 7 and 19 months of age.
(3) Exploratory: Measurement of anti-RSV antibody levels in breast milk in mothers at 1 week, 2 weeks, 4 weeks and 2 months after delivery following concurrent and sequential administration of vaccines against pertussis and RSV in pregnancy | 1 week, 2 weeks, 4 weeks and 2 months after delivery
  Anti-RSV antibody levels in breast milk of others at 1 week, 2 weeks, 4 weeks and 2 months after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa Abu-Raya, M.D., PhD, Principal Investigator — Canadian Center for Vaccinology, Dalhousie University
Locations (4):
- Canada (4):
  - Vaccine Evaluation Center, Vancouver, British Columbia
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Centre hospitalier universitaire Ste-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided